CLINICAL TRIAL: NCT06843564
Title: Enhanced Primary Care Telemedicine at Home: a Pilot Feasibility Trial
Brief Title: Remote Enhanced Assessment for Care at Home (REACH)
Acronym: REACH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Kristin Ray, Associate Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY24110038
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Common Childhood Illnesses
Keywords: Telemedicine; Telehealth; Pediatric
MeSH Terms: interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele-Device Kit Arm (Experimental): Families of 6 month old infants will receive tele-device kits that include thermometers, pulse oximeters, and tele-otoscopes and respiratory swab tests, which families will then have the option to use when they schedule telemedicine visits with their usual primary care practice.
  Interventions: Other: Remote Enhanced Assessment for Care at Home (REACH) Kit

INTERVENTIONS:
Other: Remote Enhanced Assessment for Care at Home (REACH) Kit — Families of 6 month old infants will receive tele-device kits that include thermometers, pulse oximeters, and tele-otoscopes and respiratory swab tests, which families will then have the option to use when they schedule telemedicine visits with their usual primary care practice.
  Note that the investigators are not studying the devices themselves; the investigators are instead studying health care use and experiences when these devices are made available.

SUMMARY:
The goal of this single arm pilot clinical trial is to test the feasibility and acceptability of providing families of infants with kits of tele-peripheral devices to use during telemedicine visits with their usual primary care practice.

The main question it aims to answer are:

- the feasibility of providing families of infants with a kit to tele-peripheral devices to use during at-home, same-day live-interactive primary care telemedicine visits.

Participants will receive a kit with tele-peripheral devices which they will have the option to use during telemedicine visits with their primary care practice. Participants will be asked to consent to electronic record review and to complete surveys about their experiences receiving care.

DETAILED DESCRIPTION:
The investigators will prospectively enroll 100 children (6 month 0 days to 8 months 30 days) in this one-arm pilot feasibility study. Enrolled participants will receive kits including pulse oximeters, thermometers, and tele-otoscopes as well as respiratory viral swab tests and will complete a test call with study team members to confirm ability to connect and use the devices.

After enrollment, families will continue to seek care based on their own preferences and primary care clinic guidance, but will have the ability to provide additional information to their primary care clinicians when primary care telemedicine visits occur.

The investigators will ask families to complete online surveys at 0, 30, and 180 days, and the investigators will perform chart reviews to capture visits (telemedicine and in-person to primary care, urgent care, and emergency department) and antibiotic receipt.

ELIGIBILITY:
Inclusion Criteria:

* Infants receiving care at study sites presenting for primary care child visit
* Infants between 6m0d and 20m30d

Exclusion Criteria:

* Caregiver not able to consent in English or Spanish
* Child has chronic condition (prematurity <33 weeks, congenital anomaly)
* Child is ward of the state
* Family lacks device and/or wifi plan to be able to participate in telemedicine visits

Ages: 6 Months to 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Retention | From enrollment to survey completed 6 months after enrollment, up to 18 months
  Percent who complete 6 months survey

SECONDARY OUTCOMES:
Recruitment | Day approached for recruitment, up to one year
  Percent of individuals approached who consent
Caregiver Satisfaction | From enrollment to survey completed 6 months after enrollment, up to 18 months
  Caregiver satisfaction with care using the tele-device kit as reported at 6 month survey. Satisfaction will be assessed a single Likert scale survey item, ranging from 0 to 4, with higher scores indicating greater satisfaction with care.
Kit utilization | From enrollment to survey completed 6 months after enrollment
  Number of primary care telemedicine visits where kit devices are and are not used, assessed through both survey and through chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ray, MD, MS, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Children's Hospital of Pittsburgh Primary Care Center, Pittsburgh, Pennsylvania
  - UPMC Children's Community Pediatrics - Castle Shannon, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No